CLINICAL TRIAL: NCT05852522
Title: NCT MASTER Plattform Molecularly Aided Stratification for Tumor Eradication Research
Brief Title: Molecularly Aided Stratification for Tumor Eradication Research
Acronym: NCT-MASTER
Status: Recruiting | Type: Observational
Sponsor: German Cancer Research Center (Other)
Collaborators: German Consortium for Translational Cancer Research (Other)
Responsible Party: Sponsor
Other Study IDs: TMO0001
Record Dates: First submitted 2023-04-24; First posted 2023-05-10 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-06

CONDITIONS: Rare Cancers; Multiomics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — fresh frozen tumor, DNA, RNA
Oversight: Data Monitoring Committee: Yes | US Export: No

SUMMARY:
NCT/DKFZ/DKTK MASTER is a prospective, continuously recruiting, multicenter observational study for biology-guided stratification of adults with rare cancers, including rare subtypes of common entities, using comprehensive molecular profiling, and clinical decision-making in a multidisciplinary molecular tumor board.

ELIGIBILITY:
Inclusion Criteria:

Rare cancer (Incidence <6/100,000 persons/year) or Rare subtype of a more common entity (case-by-case decision; example: pancreatic ductal adenocarcinoma without KRAS mutation)

Metastatic and/or locally advanced cancer with no curative therapy option and indication for systemic therapy

Exclusion Criteria:

Severe neurological or psychiatric disorder interfering with the ability to give oral and written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from university hospital Heidelberg and all German Consortium for Translation Research sites
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-11-11 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 5 years
  Time period of progression survival from date of multiomics analysis
overall survival | 10 years
  time period of survival from date of diagnosis

SECONDARY OUTCOMES:
response to antitumor treatment | 5 months
  response according to RECIST v.1.1 criteria to antitumor treatment applied after multiomics analysis

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Fröhling, M.D., Principal Investigator — German Cancer Research Center
Locations (1):
- German Cancer Research Center, Heidelberg, Germany

REFERENCES:
- [Background] Jahn A, Rump A, Widmann TJ, Heining C, Horak P, Hutter B, Paramasivam N, Uhrig S, Gieldon L, Drukewitz S, Kubler A, Bermudez M, Hackmann K, Porrmann J, Wagner J, Arlt M, Franke M, Fischer J, Kowalzyk Z, William D, Weth V, Oster S, Frohlich M, Hullein J, Valle Gonzalez C, Kreutzfeldt S, Mock A, Heilig CE, Lipka DB, Mohrmann L, Hanf D, Oles M, Teleanu V, Allgauer M, Ruhnke L, Kutz O, Knurr A, Lassmann A, Endris V, Neumann O, Penzel R, Beck K, Richter D, Winter U, Wolf S, Pfutze K, Georg C, Meissburger B, Buchhalter I, Augustin M, Aulitzky WE, Hohenberger P, Kroiss M, Schirmacher P, Schlenk RF, Keilholz U, Klauschen F, Folprecht G, Bauer S, Siveke JT, Brandts CH, Kindler T, Boerries M, Illert AL, von Bubnoff N, Jost PJ, Metzeler KH, Bitzer M, Schulze-Osthoff K, von Kalle C, Brors B, Stenzinger A, Weichert W, Hubschmann D, Frohling S, Glimm H, Schrock E, Klink B. Comprehensive cancer predisposition testing within the prospective MASTER trial identifies hereditary cancer patients and supports treatment decisions for rare cancers. Ann Oncol. 2022 Nov;33(11):1186-1199. doi: 10.1016/j.annonc.2022.07.008. Epub 2022 Aug 18. PMID 35988656
- [Background] Horak P, Heining C, Kreutzfeldt S, Hutter B, Mock A, Hullein J, Frohlich M, Uhrig S, Jahn A, Rump A, Gieldon L, Mohrmann L, Hanf D, Teleanu V, Heilig CE, Lipka DB, Allgauer M, Ruhnke L, Lassmann A, Endris V, Neumann O, Penzel R, Beck K, Richter D, Winter U, Wolf S, Pfutze K, Georg C, Meissburger B, Buchhalter I, Augustin M, Aulitzky WE, Hohenberger P, Kroiss M, Schirmacher P, Schlenk RF, Keilholz U, Klauschen F, Folprecht G, Bauer S, Siveke JT, Brandts CH, Kindler T, Boerries M, Illert AL, von Bubnoff N, Jost PJ, Spiekermann K, Bitzer M, Schulze-Osthoff K, von Kalle C, Klink B, Brors B, Stenzinger A, Schrock E, Hubschmann D, Weichert W, Glimm H, Frohling S. Comprehensive Genomic and Transcriptomic Analysis for Guiding Therapeutic Decisions in Patients with Rare Cancers. Cancer Discov. 2021 Nov;11(11):2780-2795. doi: 10.1158/2159-8290.CD-21-0126. Epub 2021 Jun 10. PMID 34112699
- [Background] Horak P, Klink B, Heining C, Groschel S, Hutter B, Frohlich M, Uhrig S, Hubschmann D, Schlesner M, Eils R, Richter D, Pfutze K, Georg C, Meissburger B, Wolf S, Schulz A, Penzel R, Herpel E, Kirchner M, Lier A, Endris V, Singer S, Schirmacher P, Weichert W, Stenzinger A, Schlenk RF, Schrock E, Brors B, von Kalle C, Glimm H, Frohling S. Precision oncology based on omics data: The NCT Heidelberg experience. Int J Cancer. 2017 Sep 1;141(5):877-886. doi: 10.1002/ijc.30828. Epub 2017 Jun 21. PMID 28597939